CLINICAL TRIAL: NCT05069935
Title: A Phase I, Open-Label, Multicenter Study of FT538 in Combination With Monoclonal Antibodies in Subjects With Advanced Solid Tumors
Brief Title: FT538 in Combination With Monoclonal Antibodies in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated by the Sponsor.
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FT538-102
Record Dates: First submitted 2021-09-10; First posted 2021-10-06 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Solid Tumor, Adult
Keywords: anti-PD-1 / PD-L1 antibodies approved; HER2+; Metastatic CRC; Head and Neck Squamous Cell Carcinoma; NK Cells; Urothelial Cancer; Renal Cell Carcinoma; merkel cell carcinoma; non-small cell lung cancer; NSCLC; triple negative breast cancer; immune checkpoint inhibitor; melanoma, renal cell carcinoma, lung cancer,; triple-negative breast cancer,; head and neck squamous cell carcinoma,; urothelial carcinoma (UC),; Merkel cell carcinoma, squamous; hepatocellular carcinoma; gastric cancer, esophageal cancer, endometrial cancer,
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Carcinoma, Merkel Cell; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Melanoma; Lung Neoplasms; Carcinoma, Transitional Cell; Carcinoma, Hepatocellular; Stomach Neoplasms; Esophageal Neoplasms; Endometrial Neoplasms | interventions — Cyclophosphamide; fludarabine; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): * Cohort A: FT538 plus avelumab in subjects with advanced solid tumors malignancies where anti-PD-1/PD-L1 antibodies are approved
  * Cohort B: FT538 plus trastuzumab in subjects with advanced documented HER2+ tumors
  * Cohort C: FT538 plus cetuximab in subjects with advanced colorectal cancer (CRC) or head and neck squamous cell carcinoma (HNSCC)
  Interventions: Drug: FT538; Drug: Cyclophosphamide; Drug: Fludarabine; Combination Product: Monoclonal antibody - Dose Escalation
- Dose Expansion (Experimental): * Cohort A, Arm 1: FT538 plus avelumab in subjects with advanced solid tumors malignancies where anti-PD-1/PD-L1 antibodies are approved (except urothelial carcinoma (UC))
  * Cohort A, Arm 2: FT538 plus an anti-PD-1 antibody (nivolumab or pembrolizumab) in subjects with solid tumor malignancies where anti-PD-1/PD-L1 antibodies are approved (except UC)
  * Cohort B, Arm 1: FT538 plus trastuzumab in subjects with HER2+ tumors
  * Cohort C, Arm 1: FT538 plus cetuximab in subjects with advanced CRC or HNSCC
  Subjects with UC may be enrolled in the randomized expansion cohorts as follows:
  * Cohort A, Arm R1: FT538 plus avelumab
  * Cohort A, Arm R2: FT538 plus atezolizumab
  Interventions: Drug: FT538; Drug: Cyclophosphamide; Drug: Fludarabine; Combination Product: Monoclonal antibody - Dose Expansion

INTERVENTIONS:
Drug: FT538 — FT538 is an allogeneic natural killer (NK)-cell immunotherapy
  Other Names: NK Cell Therapy
Drug: Cyclophosphamide — Lympho-conditioning agent
  Other Names: Cy
Drug: Fludarabine — Lympho-conditioning agent
  Other Names: Flu
Combination Product: Monoclonal antibody - Dose Escalation — either avelumab, trastuzumab or cetuximab
  Other Names: mAb
  Arms: Dose Escalation
Combination Product: Monoclonal antibody - Dose Expansion — either avelumab, atezolizumab, nivolumab, pembrolizumab, trastuzumab or cetuximab
  Other Names: mAb
  Arms: Dose Expansion

SUMMARY:
This is a Phase 1 dose-finding study of FT538 in combination with monoclonal antibodies.

DETAILED DESCRIPTION:
This is a Phase 1 dose-finding study of FT538 given in combination with a monoclonal antibody following lymphodepletion in subjects with advanced solid tumors. The study will consist of a dose-escalation stage and an expansion stage where participants will be enrolled into indication-specific cohorts.

ELIGIBILITY:
Inclusion Criteria:

Subjects with locally advanced or metastatic disease who have progressed after at least one line of therapy and diagnosis of one of the following by treatment cohort:

* Cohort A: The following solid tumor malignancies where anti-PD-1/PD-L1 antibodies are approved: cutaneous melanoma, non-small cell/small cell lung cancer, renal cell carcinoma, head and neck squamous cell cancer, microsatellite instability-high/ mismatch repair deficient cancer, gastric cancer, esophageal cancer, cervical cancer, merkel cell carcinoma, endometrial carcinoma, tumor mutation burden-high ≥ 10 mutations/megabase], cutaneous squamous cell carcinoma, triple-negative breast cancer.
* Cohort B: HER2+ breast cancer that has relapsed or progressed on trastuzumab and progressed on either pertuzumab or HER2-targeting antibody drug conjugate; HER2+ gastric cancer that has relapsed or progressed on trastuzumab-containing therapy; OR any other HER2+ solid tumor having progressed on at least one line of standard-of-care therapy. For any tumor type in this cohort, HER2 status must be documented by a U.S. Food and Administration (FDA) approved test to be ≥2+ IHC or Average HER2 copy number ≥4 signals per cell by in situ hybridization.
* Cohort C: CRC having progressed following prior cetuximab treatment or has KRAS/NRAS mutation; HNSCC having progressed following prior cetuximab.

Capable of giving signed informed consent

Aged ~ 18 years old

Willingness to comply with study procedures and duration

Measurable disease per RECIST v1.1

For subjects with >1 measurable lesion by RECIST v1.1 that can be safely accessed, willingness to undergo tumor biopsy

Contraceptive use for women and men as defined in the protocol

Exclusion Criteria:

Pregnant or breast-feeding women

ECOG performance status greater than or equal to 2

Evidence of insufficient organ function

Clinically significant cardiovascular disease including left-ventricular ejection fraction < 45%

Receipt of therapy within 2 weeks prior to Day 1 or five half-lives, whichever is shorter or any investigational therapy within 28 days prior to Day 1

Known active central nervous system (CNS) involvement by malignancy that hasn'thas not remained stable for at least 3 months following effective treatment for CNS disease

Non-malignant CNS disease such as stroke, epilepsy, CNS vasculitis or neurodegenerative disease or receipt of medications for these conditions

Currently receiving or likely to require immunosuppressive therapy Active bacterial, fungal, or viral infections including hep B, Hep C or HIV Live vaccine within 6 weeks prior to start of lympho-conditioning

Known allergy to albumin (human) or DMSO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Define the Recommended Phase 2 Dose (RP2D) | Up to ~1.5 years
  To define the RP2D of FT538 in combination with the following mAbs in subjects with advanced solid tumors: avelumab, trastuzumab, cetuximab, atezolizumab, nivolumab, and pembrolizumab
Incidence and Severity of Adverse Events (AEs)0 | Up to ~5 years
  To evaluate the safety and tolerability of FT538 in combination with the following mAbs in subjects with advanced solid tumors: avelumab, trastuzumab, cetuximab, atezolizumab, nivolumab, and pembrolizumab

CONTACTS AND LOCATIONS:
Overall Officials: Fate Trial Disclosure, Study Director — Fate Therapeutics
Locations (4):
- United States (4):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Sarah Cannon, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No